CLINICAL TRIAL: NCT04816227
Title: Expression Profile Study of Macrophages From Patients Affected by Amyotrophic Lateral Sclerosis (ALS) or Other Related Motor Impairments
Brief Title: Expression Profile Study of Macrophages From Patients Affected by ALS or Other Related Motor Impairments
Acronym: Mac2ALS
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C20-55; 2020-A03348-31 (Registry Identifier: ID RCB)
Record Dates: First submitted 2021-03-19; First posted 2021-03-25 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Amyotrophic Lateral Sclerosis (ALS): Blood draw
- asymptomatic carriers of ALS mutations: Blood draw
- patients with motor impairment other than ALS: Blood draw
- healthy controls: Blood draw

SUMMARY:
The aim of this project is to analyze the macrophage transcriptome and protein markers of Amyotrophic Lateral Sclerosis (ALS) patients compared to controls (non-affected individuals, patients with other motor impairments) and asymptomatic ALS gene carriers, to find new pathways for therapeutic targets and disease biomarkers.

DETAILED DESCRIPTION:
Amyotrophic Lateral Sclerosis (ALS) is the most common motor neuron disease in adults affecting upper and lower motor neurons resulting in progressive muscle atrophy and paralysis of the patients within 2 to 5 years. The majority of ALS cases are sporadic (SALS), 5 to 10% are familial forms (FALS). In France, the most frequent mutation is an intronic hexanucleotide expansion in the C9orf72 gene, representing 46% of FALS followed by mutations in the first discovered ALS gene, SOD1 accounting for around 10% of FALS. Using mutant SOD1 ALS mouse models, the investigators and others have shown that motor neurons degenerated through a non-cell autonomous mechanism involving microglial cells. Microglial cells are the macrophages of the central nervous system (CNS) capable of producing neurotrophic or neurotoxic factors. Microglial cells are part of the myeloid lineage like macrophages at the periphery, however these two cell types have different developmental origins and are in different environments. Spinal motor neurons are particular neurons since their cell body is in the CNS, and therefore surrounded by microglial cells, while their axon extends at the periphery and is therefore in contact with peripheral macrophages. The investigators have shown that (i) peripheral macrophages in affected peripheral nerves of ALS mouse models and ALS patient post-mortem tissues were activated, (ii) in ALS mouse models, both microglial cells but also peripheral macrophages participated in disease progression and (iii) peripheral macrophages were able to influence microglial cell reactivity.

The working hypothesis is that peripheral macrophages are themselves (and not just microglial cells) involved in ALS and with this project the investigators want to compare macrophages from ALS patients and controls using macrophages derived from blood monocytes. The aim is to analyze the macrophage transcriptome and protein markers of Amyotrophic Lateral Sclerosis (ALS) patients compared to controls (non-affected individuals, patients with other motor impairments) and asymptomatic ALS gene carriers, to find new pathways to target and disease biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Agree to participate in this research and have signed an informed consent
* Be able to understand the objectives and procedures of the study
* Be affiliated to French social security or equivalent
* Meet one of the criteria below:

  (i) Be affected by Amyotrophic Lateral Sclerosis (ALS) definite, probable or possible (El Escorial criteria) sporadic SALS (no known history in the family) or familial FALS (at least one other member of the family affected), (ii) not being affected by ALS but having a close relative who has or has been diagnosed with ALS and has or is a carrier of a known mutation causing ALS and has consented to a genetic analysis, (iii) Have a motor impairment including the following pathologies: Motor neuropathy, myopathy, Myositis, Spastic paraplegia, Cram / fasciculation syndrome, Chronic inflammatory polyradiculitis, somatization disorder, Anterior spinal artery syndrome, encephalitis, myelitis, Peroneal neuropathy, cervical myelopathy with radiculopathy, spinocerebellar ataxia, Kennedy disease, Spinal atrophy, Hereditary distal motor neuropathy.

(iv) be accompanying a person with ALS or other motor impairment that is followed by one of the doctors from the ALS referral center at the Pitié-Salpêtrière hospital or by a neurologist from the neurophysiology department at the Pitié-Salpêtrière hospital.

Exclusion Criteria:

* Be subjected to a legal protection measure (safeguard of justice, curatorship or guardianship)
* Refusing to participate in the study
* Whose condition, in the opinion of the doctor, is incompatible with blood draw or participation in research
* Being pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group 1: Be affected by Amyotrophic Lateral Sclerosis (ALS) definite, probable or possible (El Escorial criteria) sporadic SALS (no known history in the family) or familial FALS (at least one other member of the family affected)
  Group 2: Be a carrier of a known mutation causing ALS and be asymptomatic
  Group 3: Have a motor impairment related to ALS including the following pathologies: Motor neuropathy, myopathy, Myositis, Spastic paraplegia, Cram / fasciculation syndrome, Chronic inflammatory polyradiculitis, somatization disorder, Anterior spinal artery syndrome, encephalitis, myelitis, Peroneal neuropathy, cervical myelopathy with radiculopathy, spinocerebellar ataxia, Kennedy disease, Spinal atrophy, Hereditary distal motor neuropathy.
  Group 4: Healthy control
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2021-09-29 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Measure of transcriptome differences between the ALS group and the 3 other groups of participants. | 5 years
  Will be considered different modulation superior or equal to 1.5 fold with a statistical value of p<0.05.

CONTACTS AND LOCATIONS:
Overall Officials: François SALACHAS, MD, Study Director — APHP, Hôpital de la Salpêtrière, INSERM U1127, ICM
Locations (1):
- Département de Neurologie, Hôpital de la Pitié-Salpêtrière, Paris, France